CLINICAL TRIAL: NCT04327323
Title: Italian Registry on Cardiac Contractility Modulation Therapy
Brief Title: CCM Italian Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: S. Andrea Hospital (Other)
Collaborators: Ospedale Umberto I di Torino (Other); A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other); Ospedale Cardinal Massaia (Other); Azienda Ospedaliero Universitaria Maggiore della Carita (Other); Azienda Ospedaliera S. Maria della Misericordia (Other); IRCCS Multimedica (Other); San Giovanni di Dio Hospital (Other); Monaldi Hospital (Other); Ospedale Miulli, Acquaviva delle Fonti (Unknown); Ospedale San Bortolo di Vicenza (Other); The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other); ASST Fatebenefratelli Sacco (Other); Ospedale Policlinico San Martino (Other); Azienda Ospedaliera Bolognini di Seriate Bergamo (Other); Federico II University (Other); Ospedale Santa Croce-Carle Cuneo (Other); Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other); Martini Hospital, Turin, Italy (Other); Ospedale di Ariano Irpino (Unknown); Ospedale di Borgomanero (Unknown); ASL Verbano Cusio Ossola (Other Government); Policlinico Hospital (Other); Azienda Ospedaliero Universitaria di Cagliari (Other); Fatebenefratelli Hospital (Other); Centro Cuore Morgagni, Pedara (Unknown); Santa Maria delle Grazie Hospital (Other); Ospedale di Gorizia (Unknown); ASP Enna (Unknown); Ospedale Garibaldi, Catania (Unknown); Ospedali Riuniti Anzio-Nettuno (Unknown); Ospedale Fracastoro, Soave San Bonifacio (Unknown); Ospedale Magalini, Villafranca (Unknown); Casa di Cura Pierangeli, Pescara (Unknown)
Responsible Party: Principal Investigator, Mario Matta, M.D., S. Andrea Hospital
Other Study IDs: CCM-REG-IT
Record Dates: First submitted 2020-03-25; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure
Keywords: cardiac contractility modulation; heart failure; hospitalizations; exercise tolerance
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CCM device implantation — CCM implantation involves the introduction of two active fixation stimulation leads, fixed on the interventricular septum, and connected to the CCM generator (Optimizer Smart IV, Impulse Dynamic, and any subsequent versions of the same device) inserted in the subcutaneous or submuscular pocket. The implantation is ususally performed using vascular access via right or left cephalic or subclavian vein. The CCM signal consists of 2-3 biphasic pulses lasting 10 msec (total duration of about 20 ms) with an amplitude between 4.0 and 7.5 V, delivered during the absolute refractory period of the ventricle, at a distance of 40 msec from ventricular sensing. The CCM device is compatible with other pacing and defibrillation devices already implanted in the patient; at the time of the implantation, the devices are checked in order to confirm the absence of interference between the devices. The patient is instructed to charge the device battery weekly.

SUMMARY:
The Cardiac Contractility Modulation (CCM) system is a cardiac implantable device indicated for the treatment of patients with symptomatic heart failure with left ventricular systolic dysfunction despite optimal medical and electrical therapy. This system consists of a generator to which two stimulation leads are connected, which are fixed on the interventricular septum and deliver non-excitatory electrical signals during the absolute ventricular refractory period, with the aim of influencing the contractility properties of the myocardium in patients with chronic heart failure. Clinical data indicate that CCM therapy is safe and effective for the treatment of patients with symptomatic heart failure with reduced left ventricular systolic function, in which a significant improvement in quality of life and exercise tolerance has been shown, together with an impact on hospitalizations for heart failure.

This prospective registry includes patients undergoing CCM implantation for the above clinical indications. The inclusion criteria are age over 18; chronic heart failure with reduced left ventricular systolic function (FE ≤ 45%), symptomatic (class NYHA II or greater; class III or greater or II with episodes of acute decompensation for patients with FE 36-45%); presence of appropriate and optimized medical therapy (including beta-blockers and angiotensin-converting enzyme inhibitors or angiotensin-receptor blockers or angiotensin-receptor neprylysin inhibitors and anti-aldosterone agents); narrow QRS (<120 msec) or cardiac resynchronization therapy non-responders; written informed consent for enrollment and participation in the prospective register; life expectancy> 1 year due to the absence of non-cardiac comorbidities that reduce its prognosis; availability of venous access that can be used for the implant. The exclusion criteria are the absence of venous access available for the implant; contraindication to the interventional CCM implant procedure; life expectancy of less than one year due to non-cardiovascular comorbidities.

The aim of this multicenter, prospective, observational registry is to investigate the impact of CCM on the medium and long-term on clinical and functional characteristics of the enrolled patients at the end of the follow-up, with respect to the baseline value: NYHA class, 6-minute walk test, ejection fraction and volumes of the left ventricle, quality of life expressed through a specific questionnaire (Minnesota Living With Heart Failure Questionnaire, MLWHF), hospitalizations for heart failure or progression of the underlying heart disease. In addition, the survival of patients undergoing CCM device implantation will be assessed in an observational manner at 24 months and then annually.

In addition, adverse events related to the device implantation procedure or to CCM therapy are collected in the registry as a safety parameter. In the case of patients undergoing heart transplantation or LVAD implantation, or in the event of interruption of therapy or explantation of a device, the information will be recorded with the motivation for discontinuing treatment.

Clinical follow-up includes follow-up assessments at 3 months, 6 months, 12 months and every 6 months thereafter. Each clinical follow-up visit includes objective examination, ECG, device function check, administration of an MLWHF quality of life questionnaire, a 6-minute walk test (or cardiopulmonary exercise test) and pharmacological therapy assessment and optimization. Furthermore, during the follow-up visits at 3 months, 12 months and every 12 months thereafter, a transthoracic echocardiogram and blood chemistry tests are scheduled.

This multicenter observational prospective registry therefore aims to assess the long-term clinical impact of CCM in patients suffering from symptomatic heart failure with moderately or severely impaired systolic function. In particular, it will allow to evaluate the impact on functional capacity, symptoms and quality of life, hospitalizations, survival and device-related complications, with the aim of defining the role of CCM therapy in management of patient with heart failure with reduced left ventricular systolic function.

DETAILED DESCRIPTION:
Introduction The Cardiac Contractility Modulation (CCM) system is a cardiac implantable device indicated for the treatment of patients with symptomatic heart failure with left ventricular systolic dysfunction despite optimal medical and electrical therapy.

This system consists of a generator to which two stimulation leads are connected, which are fixed on the interventricular septum and deliver non-excitatory electrical signals during the absolute ventricular refractory period, with the aim of influencing the contractility properties of the myocardium in patients with chronic heart failure. The generator of the device is rechargeable, and the patient is equipped with a special charger, while the device can be interrogated through a special programmer.

Currently available studies indicate that CCM therapy is safe and effective for the treatment of patients with symptomatic heart failure with reduced left ventricular systolic function despite appropriate and optimized medical therapy. Based on data available from clinical studies, the application of CCM signals to the heart during the absolute refractory period can increase the contraction force of the myocardium. In particular, a significant improvement in quality of life and exercise tolerance has been reported (highlighted by the improvements in the 6-minute walking test and in the peak of VO2 in the cardiopulmonary exercise test), together with a potential impact on hospitalizations for heart failure and survival. In addition, CCM therapy reverses the characteristics of left ventricular remodeling typical of decompensation and improves left ventricular contractile reserve. These effects are the result of a chain of intracellular molecular processes, some of which become evident within a few seconds after starting the CCM. For example, CCM signals have been shown to normalize the phosphorylation of regulatory proteins such as phospholamban in vitro within a few seconds of treatment. This rapid effect triggers a series of molecular events which result in the restoration of cellular function and in the acute improvement of contractile force. On the long term, there is a progressive normalization of the abnormal expression of the fetal gene program characteristic of heart failure and a progressive reduction of the end-diastolic volume with an increase in the ejection fraction of the left ventricle. These effects on intracellular signaling mechanisms also extend to regions of the ventricle far from the impulse delivery area.

The prospective register This prospective registry includes patients undergoing CCM implantation for the presence of heart failure with reduced left ventricular systolic function (EF < 45%) who are symptomatic despite optimal pharmacological and electrical therapy. The clinical trial study (prospective registry) will be conducted in accordance with this protocol, with the Helsinki Declaration and with the favorable opinion of the local Ethics Committee of the participating Centers Full detailed inclusion and exclusion criteria are reported in the specific section.

Aim of the study This prospective observational register is intended to collect data uniformly on patients treated with CCM. The data will be used to evaluate the medium and long-term clinical and instrumental effects on patients treated with CCM therapy and will have a purely scientific value.

In particular, the objective of the registry is to investigate the impact of the CCM on the clinical and functional characteristics of the patients enrolled at the end of the follow-up with respect to the baseline value: NYHA class, 6-minute walking test distance, left ventricular ejection fraction and volumes , quality of life expressed through a specific questionnaire (Minnesota Living With Heart Failure Questionnaire, MLWHF), hospitalizations for heart failure or progression of the underlying heart disease. These parameters will be assessed and analyzed in an observational manner 24 months after the start of the study and subsequently annually.

In addition, the survival of patients undergoing CCM device implantation will be assessed in an observational manner. Finally, device-related complications will be assessed a safety outcome, and other cardiovascular adverse event will be assessed as well.

These parameters will be assessed globally in the entire enrolled population, and also separately in three pre-specified groups: patients with EF between 36% and 45% (in NYHA class III, IV or II with previous hospitalizations for heart failure); patients with EF between 25% and 36% carriers of CRT-D / P ("non-responders"); patients with EF between 25% and 35% not carriers of CRT-D / P; patients with EF <25%.

Clinical and instrumental parameters

The following data will be collected in basal conditions upon enrollment:

1. Age, gender, weight, BMI
2. Comorbidity: diabetes mellitus, hypertension, renal failure, COPD, atrial fibrillation, previous stroke, peripheral vascular disease
3. NYHA class
4. Left ventricular ejection fraction, end-systolic and end-diastolic volumes and diameters, diastolic function, degree of mitral insufficiency, right ventricle size and contractility, sPAP (echocardiogram)
5. Systolic blood pressure
6. Etiology of cardiomyopathy (ischemic, idiopathic, valvular, hypertensive, other)
7. Baseline QRS duration
8. Laboratory data (according to the normal clinical practice of the Center for heart failure patients):

   to. Hemoglobin [g / dL] b. Lymphocytes [%] c. Uric acid [mg / dL] d. Creatinine [mg / dL] e. Total cholesterol [mg / dl] f. Sodium [mmol / L] g. BNP or NT-proBNP [pg / mL] h. Soluble ST2 [ng / ml]
9. Current therapy, including the following:

   to. ACE inhibitors [Y / N] b. Beta blockers [Y / N] c. Angiotensin-receptor blockers [Y / N] d. Angiotensin-receptor neprylysin inhibitors [Y/N] e. Statins [Y / N] f. Allopurinol [Y / N] g. Aldosterone antagonists [Y / N] h. Diuretics [Y / N and dosage]
10. Previous Levosimendan cycles (number)
11. Devices already implanted before enrollment [none / CRT-P / ICD / CRT-D)
12. Number of heart failure hospitalizations in the past year
13. Quality of life, as assessed by the "Minnesota Living with Heart Failure Questionnaire" (MLWHFQ)
14. Exercise tolerance, measured with (according to the Centre's clinical practice):

    1. peak of oxygen consumption (VO 2) determined during cardiopulmonary exercise tests;
    2. 6-minute walking test distance.

Safety measures:

Adverse events related to the device, implant procedure or CCM therapy are collected in the registry as safety parameter. Each type of complication is entered in the register, classified as major if it leads to death, endangers life or requires invasive treatment, hospitalization or prolonged hospitalization due to the need to resolve the complication. The other complications are classified as minor.

In case of patients undergoing heart transplantation or LVAD implantation, or in the event of interruption of therapy or explantation of a device, the information will be recorded with the motivation for discontinuing treatment.

Device parameters

The following parameters of the CCM device will be recorded at each follow-up visit, carried out according to normal clinical practice for patients with this device:

* Stimulation activity: RV [Active / Inactive], LS [Active / Inactive]
* Amplitude of CCM stimulation [Volt] Device sensing [RV and LS]
* Percentage of CCM Therapy (i.e. percentage of heart beats that actually receive CCM therapy within the scheduled hours)
* Number of CCM therapy hours scheduled per day
* Number of actual CCM therapy hours per day

Study design This registry is a multicenter, prospective, observational, open-label study, with the aim of evaluating the clinical effect of CCM therapy during a follow-up in an open number of subjects with heart failure and moderate-to-severe left ventricular systolic dysfunction despite appropriate medical therapy, during the long term and within a minimum duration of 24 months.

The sample size is open, being an observational registry; however, a sample size of 200 pazients in anticipated to complete the enrollment and analyze the whole data; a preliminary analysis will be performed following the first 100 enrolled patients.

The implant procedure involves the introduction of two active fixation stimulation leads, fixed on the interventricular septum, and connected to the CCM generator (Optimizer Smart IV, Impulse Dynamic, and any subsequent versions of the same device) inserted in the subcutaneous or submuscular pocket. The implantation uses a vascular access via right or left cephalic or subclavian vein. The CCM signal delivered consists of 2-3 biphasic pulses lasting 10 msec (total duration of about 20 ms) with an amplitude between 4.0 and 7.5 V, delivered during the absolute refractory period of the ventricle, at a distance of 40 msec from ventricular sensing (Kuschyk J, Rev Cardiovasc Med 2017). The CCM device is compatible with other pacing and defibrillation devices already implanted in the patient; at the time of the implantation, the devices are checked in order to confirm the absence of interference between the devices. The patient is instructed to charge the device battery weekly.

Follow-up Clinical follow-up includes check-ups at 3 months, 6 months, 12 months and every 6 months thereafter.

Each clinical follow-up visit includes the execution of objective examination, ECG, control of the functioning of the device, administration of MLWHF questionnaire on quality of life, 6-minute walking test (or cardiopulmonary exercise test when required) and evaluation and titration of the pharmacological therapy.

In addition, during the 3-month, 12-month and every 12-month follow-up visits, a transthoracic echocardiogram and blood chemistry tests are scheduled.

The following data will be recorded and entered in the study database at the time of enrollment and during the follow-up visits, as per study design:

* Clinical history, including demographics and ongoing therapy
* ECG (rhythm, QRS duration)
* NYHA class
* MLWHF questionnaire score
* Six-minute walking test distance

  - Cardiopulmonary stress test results (when performed)
* Echocardiographic data (diameters and volumes of the left ventricle, left ventricular ejection fraction, diastolic function, degree of mitral insufficiency, size and contractility of the right ventricle, sPAP)
* Parameters required for calculating the SHFM score
* Device operating and programming parameters
* Pharmacological therapy during the follow-up
* Any hospitalizations for heart failure or progression of the underlying heart disease
* Administration of levosimendan
* NT-proBNP and sST2 dosage
* Possible interruption of treatment and reason for interruption
* Complications related to CCM therapy

The study does not include the execution of additional clinical investigations, instrumental examinations, administration of drugs or additional services that are not included in the normal clinical practice of the follow-up management of patients undergoing CCM therapy. The enrollment or not in the registry does not affect the indication to the device implantation, nor the management of the follow-up from a clinical-instrumental point of view or the follow-up visits. No additional expenses are foreseen by the participating centers, nor funding is expected by external companies, or compensation to the investigators or to enrolled patients. The consent or refusal to be enrolled in the registry does not alter the normal clinical management of patients undergoing CCM implantation or the treatment of heart failure.

Conclusion This multicenter observational prospective registry aims to assess the clinical impact of cardiac contractility modulation therapy (CCM) in patients with symptomatic heart failure with moderately or severely impaired left ventricular systolic function. This study will allow to evaluate the long-term clinical impact of CCM therapy on patients' functional capacity, symptoms and quality of life, hospitalizations for decompensation and progression of the underlying disease, as well as the survival and complications observed, with the objective to define the role of CCM therapy in the management of patient with heart failure with reduced left ventricular systolic function.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure with reduced left ventricular systolic function (EF ≤ 45%), symptomatic (class NYHA III or greater; or class II with previous episodes of acute decompensation for patients with FE 36-45%);
* presence of appropriate and optimized medical therapy, including: beta-blocker and angiotensin-converting enzyme inhibitor or angiotensin-receptor blocker or angiotensin-receptor neprylysin inhibitor and anti-aldosterone agent, titrated as tolerated by the patients;
* narrow QRS (<120 msec) or cardiac resynchronization carriers with documented non-response to this treatment;
* age above 18 years;
* written informed consent for enrollment and participation in the prospective register.

Exclusion Criteria:

* life expectancy < 1 year due to non-cardiac comorbidities that reduce the prognosis;
* absence of vascular access that can be used for the implant;
* other contraindications to the CCM implantation procedure (e.g. active infective processes, active severe coagulopathies);
* refusal to be enrolled in the registry.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective registry includes patients undergoing CCM implantation for the presence of symptomatic heart failure with moderately-to-severely reduced left ventricular systolic function despite optimal pharmacological and electrical therapy. The clinical trial study (prospective registry) will be conducted in accordance with this protocol, with the Helsinki Declaration and with the favorable opinion of the local Ethics Committee of the participating Centers.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Exercise tolerance | 24 months
  6-minute walking test distance (meters)
Quality of life measured by Minnesota Living With Heart Failure questionnaire | 24 months
  Minnesota Living With Heart Failure questionnaire score (scale 0-105; high scorse mean worse outcome)
Functional class | 24 months
  NYHA (New York Heart Association) class (range I-IV; IV means worse outcome)

SECONDARY OUTCOMES:
Left ventricular systolic function | 24 months
  Left ventricular ejection fraction (%)
Hospitalizations | 24 months
  hospitalizations for worsening heart failure or cardiomyopathy progression (n)
Left ventricular volume | 24 months
  Left ventricular end-systolic volume (ml)

OTHER OUTCOMES:
Survival | 24 months
  Survival (both overall and non-cardiovascular death)
Complications | 24 months
  Device-related complications
Others | 24 months
  Any cardiovascular adverse events (death, stroke, myocardial infarction, major bleedings, life-threatening ventricular arrhythmias)

CONTACTS AND LOCATIONS:
Locations (1):
- Sant'Andrea Hospital, Vercelli, VC, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borggrefe MM, Lawo T, Butter C, Schmidinger H, Lunati M, Pieske B, Misier AR, Curnis A, Bocker D, Remppis A, Kautzner J, Stuhlinger M, Leclerq C, Taborsky M, Frigerio M, Parides M, Burkhoff D, Hindricks G. Randomized, double blind study of non-excitatory, cardiac contractility modulation electrical impulses for symptomatic heart failure. Eur Heart J. 2008 Apr;29(8):1019-28. doi: 10.1093/eurheartj/ehn020. Epub 2008 Feb 12. PMID 18270213
- [Background] Kuck KH, Bordachar P, Borggrefe M, Boriani G, Burri H, Leyva F, Schauerte P, Theuns D, Thibault B; Document Reviewers; Kirchhof P, Hasenfuss G, Dickstein K, Leclercq C, Linde C, Tavazzi L, Ruschitzka F. New devices in heart failure: an European Heart Rhythm Association report: developed by the European Heart Rhythm Association; endorsed by the Heart Failure Association. Europace. 2014 Jan;16(1):109-28. doi: 10.1093/europace/eut311. Epub 2013 Nov 20. PMID 24265466
- [Background] Abraham WT, Kuck KH, Goldsmith RL, Lindenfeld J, Reddy VY, Carson PE, Mann DL, Saville B, Parise H, Chan R, Wiegn P, Hastings JL, Kaplan AJ, Edelmann F, Luthje L, Kahwash R, Tomassoni GF, Gutterman DD, Stagg A, Burkhoff D, Hasenfuss G. A Randomized Controlled Trial to Evaluate the Safety and Efficacy of Cardiac Contractility Modulation. JACC Heart Fail. 2018 Oct;6(10):874-883. doi: 10.1016/j.jchf.2018.04.010. Epub 2018 May 10. PMID 29754812
- [Background] Kloppe A, Lawo T, Mijic D, Schiedat F, Muegge A, Lemke B. Long-term survival with Cardiac Contractility Modulation in patients with NYHA II or III symptoms and normal QRS duration. Int J Cardiol. 2016 Apr 15;209:291-5. doi: 10.1016/j.ijcard.2016.02.001. Epub 2016 Feb 3. PMID 26908357
- [Background] Kuschyk J, Roeger S, Schneider R, Streitner F, Stach K, Rudic B, Weiss C, Schimpf R, Papavasilliu T, Rousso B, Burkhoff D, Borggrefe M. Efficacy and survival in patients with cardiac contractility modulation: long-term single center experience in 81 patients. Int J Cardiol. 2015 Mar 15;183:76-81. doi: 10.1016/j.ijcard.2014.12.178. Epub 2015 Jan 20. PMID 25662055
- [Background] Butter C, Rastogi S, Minden HH, Meyhofer J, Burkhoff D, Sabbah HN. Cardiac contractility modulation electrical signals improve myocardial gene expression in patients with heart failure. J Am Coll Cardiol. 2008 May 6;51(18):1784-9. doi: 10.1016/j.jacc.2008.01.036. PMID 18452785
- [Background] Imai M, Rastogi S, Gupta RC, Mishra S, Sharov VG, Stanley WC, Mika Y, Rousso B, Burkhoff D, Ben-Haim S, Sabbah HN. Therapy with cardiac contractility modulation electrical signals improves left ventricular function and remodeling in dogs with chronic heart failure. J Am Coll Cardiol. 2007 May 29;49(21):2120-8. doi: 10.1016/j.jacc.2006.10.082. Epub 2007 May 17. PMID 17531662
- [Background] Anker SD, Borggrefe M, Neuser H, Ohlow MA, Roger S, Goette A, Remppis BA, Kuck KH, Najarian KB, Gutterman DD, Rousso B, Burkhoff D, Hasenfuss G. Cardiac contractility modulation improves long-term survival and hospitalizations in heart failure with reduced ejection fraction. Eur J Heart Fail. 2019 Sep;21(9):1103-1113. doi: 10.1002/ejhf.1374. Epub 2019 Jan 16. PMID 30652394